CLINICAL TRIAL: NCT00905801
Title: CTP (Computed Tomography Perfusion) Imaging of Lung Cancer
Brief Title: Computed Tomography (CT) Perfusion Imaging of Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-PI left institution, PI not pursuing
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-149
Record Dates: First submitted 2009-05-15; First posted 2009-05-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma, Non Small Cell Lung
Keywords: Non small cell lung cancer; NSCLC; CTP; Perfusion; Imaging
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A CT Perfusion (Other): Arm A Procedure
  On the first required study visit, subject will undergo one SOC CT scan followed by the research component:
  * CTP imaging: Single bed position CTP examination, which includes injection of 30 cc of contrast agent, over the predetermined lesion from clinical scan
  * Subject will stand up and walk around, and then lay back down
  * CT Perfusion imaging: Second single bed position CTP examination, which includes injection of 30 cc of contrast agent, over the predetermined lesion from their clinical scan
  Procedures will be repeated at optional second study visit ~6-8 weeks later.
  Interventions: Other: CT Perfusion
- Arm B CT Perfusion (Other): Arm B Procedure
  On the first required study visit, subject will undergo one SOC CT scan followed by the research component:
  - CT Perfusion imaging: Single bed position CTP examination, which includes injection of 30 cc of contrast agent, over the predetermined lesion from clinical scan
  Procedures will be repeated at optional second study visit ~6-8 weeks later.
  Interventions: Other: CT Perfusion

INTERVENTIONS:
Other: CT Perfusion — Subjects will be examined with a CTP Imaging protocol which comprises repeated CT-scans of the tumor over a period of 50 seconds following the injection of a 30cc bolus of an FDA-approved low osmolar, iodinated CT contrast agent using a 64 row-multidetector row CT unit (LightSpeed VCT, GE Healthcare, Milwaukee, WI). One scan will be acquired every 3 seconds over a 50s period at 100 kV, and 100mA tube current. With this method, a 4cm long segment of the tumor can be analyzed, and 32 images of a slice thickness of 1.25 mm reconstructed simultaneously. Images will be evaluated using standard CT blood flow software (Perfusion 2, AW, GE Health Care, Milwaukee, WI).

SUMMARY:
This is an experimental study of the feasibility and efficacy of CT perfusion (CTP) imaging (CT blood flow measurements) in subjects with non-small cell lung cancer.

DETAILED DESCRIPTION:
Drug/Device Information

1) Contrast

30 cc bolus of a low osmolar, iodinated CT contrast agent, which is FDA approved and used in the clinical CT Imaging procedure.

2) Scanner

The 64 row-multidetector row CT unit (LightSpeed VCT, GE Healthcare, Milwaukee, WI) is FDA approved for clinical CT imaging

Research Design and Methods

1) Primary Endpoint

1. Diagnostic yield of tumor perfusion measurements using a contrast assisted computed tomography technique.

2) Secondary Endpoints

1. Reproducibility of tumor blood flow estimates derived by CT.
2. Assessment of the association between tumor vascularity responses after two cycles of chemotherapy and subsequent best tumor response according to standard anatomic response evaluation criteria (RECIST).
3. Predictive value of tumor blood flow for patient survival, compared to the predictive power of tumor size determinations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with any stage non-small cell lung cancer (NSCLC) who will undergo imaging with CT of the chest with intravenous contrast as standard of care. Other imaging tests will be performed as clinically indicated.
* Patient should be receiving, or planning to receive, or have received systemic therapy (chemotherapy and/or novel agents) treatment with or without radiotherapy. Patients should not be receiving adjuvant or postoperative treatment but neoadjuvant treatment is allowed.
* Histologically or cytologically proven NSCLC.
* At least one measurable primary or other intrathoracic/supraclavicular lesion ≥ 1 cm, according to Response Evaluation Criteria in Solid Tumors (RECIST); this lesion should be either proven to be malignant by biopsy or be considered malignant based on its evolution on previous imaging studies. A scan within 3-6 months prior to registration can be used as the baseline scan.
* Age 18 years or older and ability to provide informed consent.
* Subjects must use medically appropriate contraception if sexually active; women of childbearing potential must not be pregnant or breastfeeding
* Subjects must have normal renal function to participate. Standard laboratory testing to evaluate renal function will be performed prior to administering IV contrast and will be available as standard of care. Renal impairment is defined as a glomerular filtration rate of less than 60 ml/min/1.73 m2 BSA, derived from the patients' serum creatinine concentration.

Exclusion Criteria:

* Subjects of reproductive potential, who are sexually active but unwilling and/or unable to use medically appropriate contraception, or women who are pregnant or breastfeeding;
* Established allergy to iodine containing contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of tumor perfusion measurements using a contrast assisted computed tomography technique. | Data collected during one required study visit, and optional second study visit ~6-8 weeks later.

SECONDARY OUTCOMES:
Reproducibility of tumor blood flow estimates derived by CT. | Data collected during one required study visit, and optional second study visit ~6-8 weeks later.
Assessment of the association between tumor vascularity responses after two cycles of chemotherapy and subsequent best tumor response according to standard anatomic response evaluation criteria (RECIST). | Data collected during one required study visit, and optional second study visit ~6-8 weeks later.
Predictive value of tumor blood flow for patient survival, compared to the predictive power of tumor size determinations. | Data collected during one required study visit, and optional second study visit ~6-8 weeks later; and during SOC follow-up for survival.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Socinski, MD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Hillman Cancer Center: University of Pittsburgh Cancer Institute / UPMC Department of Radiology, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania